CLINICAL TRIAL: NCT02919813
Title: Mindfulness-Based Group Cognitive Behavior Therapy for Women With Provoked Localized Vulvodynia: A Randomized Pilot Study
Brief Title: M-gCBT for Women With Provoked Localized Vulvodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Catherine M Leclair, MD, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OHSU IRB 15221
Record Dates: First submitted 2016-07-19; First posted 2016-09-29 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2019-12

CONDITIONS: Provoked Localized Vulvodynia
Keywords: mindfulness group therapy; vulvodynia; vulvar pain
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- M-gCBT Group (Active Comparator): Mindfulness Based Group Cognitive Behavior Therapy (M-gCBT Group) is a type of counseling that teaches women to have more control over their pain.
  Interventions: Behavioral: Mindfulness Based Group Cognitive BehaviorTherapy
- Educational Seminars (Active Comparator): Educational seminars teach women about the different aspects of PLV that affect emotional and physical health.
  Interventions: Behavioral: Educational Seminars

INTERVENTIONS:
Behavioral: Mindfulness Based Group Cognitive BehaviorTherapy — Mindfulness Based Group Cognitive Behavior Therapy is a type of counseling that teaches women to have more control over their pain.
  Other Names: M-gCBT
  Arms: M-gCBT Group
Behavioral: Educational Seminars — Educational seminars teach women about the different aspects of PLV that affect emotional and physical health.
  Arms: Educational Seminars

SUMMARY:
The purpose of this study is to learn more about Mindfulness based Group Cognitive Behavior Therapy (M-gCBT) as a treatment for Provoked Localized Vulvodynia (PLV). M-gCBT is a counseling technique that has been shown to reduce pain and anxiety with other medical conditions, including chronic pain conditions. The investigators wish to see if participation in M-gCBT course will help reduce anxiety, fear, and pain in women with PLV greater than education alone. Both techniques use a group setting including other women with PLV. "Mindfulness-Based Group Cognitive Behavior Therapy for Women with Localized Vulvodynia" is a study designed to learn more about the use of mindfulness based group cognitive behavior therapy for PLV pain and anxiety over education alone. Participants will be randomized to one of two groups: mindfulness based cognitive behavior therapy or group education seminars.

DETAILED DESCRIPTION:
M-gCBT is a type of counseling that teaches women to have more control over their pain. Educational seminars teach women about the different aspects of PLV that affect emotional and physical health. Both groups will be given a binder containing course material at the first session and homework at each session that you will be asked to complete. The group education seminars will include an informational video clip reviewing an aspect of PLV and sexuality and will be followed by a group discussion facilitated by an instructor. Each session will involve a teacher and a small group of 6 to 12 women with PLV. Additionally, women in both groups will be asked to perform a weekly test to measure pain and to complete a daily diary.

ELIGIBILITY:
Inclusion Criteria:

1. Reported dyspareunia for at least 6 months in non-pregnant, healthy women over aged 18-45 years old meeting Friedrich's criteria for PLV.51
2. Qtip Test51-52, 54 mean verbal rating score of ≥4/10 in 4 of 6 defined points of the vestibule (2, 4, 6, 8, 10, 12 o'clock), and have received a Qtip Test score of verbal ≤ 2/10 for the labia majora and minora, intra labial sulcus, and perineum.
3. Ability to insert a regular Tampax® tampon
4. Baseline tampon test pain score ≥80mm
5. Phone access
6. Lives within 60 miles with reliable transportation

Exclusion Criteria:

1. Pregnancy
2. Active counseling or mindfulness training (within 6 months of study)
3. Any other clinical reason for dyspareunia (endometriosis pain, chronic pelvic pain, vulvar dermatoses such as psoriasis, lichen sclerosus, etc).
4. Impaired cognition or disruptive behavior not conducive to group dynamic
5. Planned long term travel or surgery during study period
6. Unable or unwilling to complete baseline assessments or agree to be randomized.
7. Axis 2 diagnosis, chronic substance abuse, suicidality or disruptive to group dynamic
8. Non-English speaking

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Leclair, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | M-gCBT Group | Educational Seminars
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M-gCBT Group | Educational Seminars | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (6.2) | 29.1 (6.1) | 31.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 11 | 16 | 27
  Race: Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 17 | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.5 (5.3) | 22.1 (3.2) | 22.3 (4.2)
Relationship status [Count of Participants; unit: Participants]
  Partnered | 12 | 13 | 25
  Not partnered | 2 | 4 | 6
Previous physical therapy [Count of Participants; unit: Participants] | 10 | 15 | 25
Previous counseling [Count of Participants; unit: Participants] | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Tampon Test
Description: The change from baseline in pain measured by the Tampon Test at 6 months. The tampon test is a validated tool used to measure (vulva) vestibular skin pain by having participants insert and remove a tampon. Participants will be asked to rate their pain along a 100 mm Visual Analog Scale on a scale of 0 (No pain) to 10 (Pain as bad as you can imagine). This test will occur at baseline and 6 months follow up.
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
units on a scale | -2.43 [-3.41 to -1.46] | -1.88 [-2.83 to -0.92]

2. Secondary Outcome: Sexual Distress Survey Response
Description: Change from baseline in sexual distress at 6 months. Participants will complete a Female Sexual Distress Scale (FSDS) survey to rate their feelings associated with sexual activities; range 0 (better outcome) - 52 (worse outcome). The FSDS surveys will be completed at baseline and 6 months follow up. A negative change in FSDS score from baseline indicates less sexual distress over time (better outcome) and a positive change in FSDS score from baseline indicates more sexual distress over time (worse outcome).
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
score on a scale | -14.53 [-20.09 to -8.98] | -10.52 [-15.39 to -5.65]

3. Secondary Outcome: Sexual Function Questionnaire Response
Description: Change from baseline in sexual function at 6 months. Participants will complete a Female Sexual Function Index (FSFI) survey which asks questions about participants sexual feelings over the past 4 weeks; range 2 (worse outcome) - 95 (better outcome). The FSFI surveys will be completed at baseline and 6 months follow up. A negative change in FSFI score from baseline indicates less sexual function over time (worse outcome) and a positive change in FSFI score from baseline indicates more sexual function over time (better outcome).
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
score on a scale | 13.33 [4.14 to 22.52] | 1.23 [-6.40 to 8.87]

4. Secondary Outcome: Depression Questionnaire Response
Description: Change from baseline in depression at 6 months. Participants will complete the Beck Depression Inventory (BDI-PC) questionnaire, which consists of 21 groups of statements where participants selects which statement best describes how they have been feeling during the past 2 weeks. Total score = sum of 21 statement subscales; range 0 (better outcome) - 63 (worse outcome). The BDI-PC surveys will be completed at baseline and 6 months follow up. A negative change in BDI-PC score from baseline indicates less depression over time (better outcome) and a positive change in BDI-PC score from baseline indicates more depression over time (worse outcome).
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
score on a scale | -5.03 [-8.49 to -1.56] | -0.02 [-3.27 to 3.23]

5. Secondary Outcome: Anxiety Questionnaire Response
Description: Change from baseline in anxiety at 6 months. Participants will complete the General Anxiety Disorder-7 (GAD-7) scale questionnaire. The GAD-7 consists of 7 problems where participants rate how often they have been bothered by those problems during the past 2 weeks. Total score = sum of 7 subscales; range 0 (better outcome) - 21 (worse outcome). The GAD-7 surveys will be completed at baseline and 6 months follow up. A negative change in GAD-7 score from baseline indicates less anxiety over time (better outcome) and a positive change in GAD-7 score from baseline indicates more anxiety over time (worse outcome).
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
score on a scale | -3.10 [-4.89 to -1.31] | -0.26 [-1.86 to 1.33]

6. Secondary Outcome: Pain Catastrophizing Scale Response
Description: Change from baseline in pain catastrophizing at 6 months. Participants will complete the Pain Catastrophizing Scale survey. The survey consists of thirteen statements describing different thoughts and feelings that may be associated with pain. Total score = sum of 13 statement subscales; range 0 (better outcome) - 52 (worse outcome). The pain catastrophizing surveys will be completed at baseline and 6 months follow up. A negative change in score from baseline indicates less pain catastrophizing over time (better outcome) and a positive change in score from baseline indicates more pain catastrophizing over time (worse outcome).
Time Frame: Change from time of enrollment until 6 months after study
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 14 | 17
score on a scale | -12.24 [-17.37 to -7.11] | -11.16 [-15.67 to -6.66]

7. Secondary Outcome: Quality of Life Questionnaire Response
Description: Perceived treatment improvement and satisfaction in quality of life questionnaire. Questionnaires for quality of life at end of group intervention and at 3 months and 6 months follow up.
Time Frame: Change from end of study until 6 months after study
Population: Outcome was not analyzed.
Arm/Group | M-gCBT Group | Educational Seminars
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Per protocol, Adverse Event data were not collected for this study
Description: Per protocol, Adverse Event data were not collected for this study
Arm/Group | M-gCBT Group | Educational Seminars
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT02919813/Prot_SAP_000.pdf